CLINICAL TRIAL: NCT02801695
Title: Evaluation of the Efficacy of Citrulline Supplementation on the Delay of Delivery for Women Hospitalized for Pre-eclampsia (CITRUPE)
Acronym: CITRUPE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC15_0475
Record Dates: First submitted 2016-06-03; First posted 2016-06-16 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Pre-eclampsia; Pregnancy
Keywords: pre-eclampsia; citrulline; pregnancy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Citrulline (Experimental): Bolus (9g) after patient stabilization, then 3g 3 times a day until delivery
  Interventions: Drug: Citrulline
- Lactose (Placebo Comparator): Bolus (9g) after patient stabilization, then 3g 3 times a day until delivery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citrulline — Citrulline supplementation
  Arms: L-Citrulline
Drug: Placebo — Placebo
  Arms: Lactose

SUMMARY:
Pre-eclampsia (PE) complicates 2-8 % of pregnancies and is associated with high maternal and fetal morbidity and mortality. The early clinical manifestations are the occurrence of a maternal blood pressure and proteinuria. Placental dysfunction impairs the nutrient supply to the fetus, and may be the cause of an intrauterine growth retardation (IUGR). This is a disease that causes prematurity and currently the only known cure is delivery of the placenta. Nitrogen monoxide (NO) regulates the placental blood flow. However, pre-eclampsia is directly related to a failure of placental NO production. In this context, several clinical trials have tested the effect of NO donors such as L- arginine. However, supplementation with L -Arginine in a randomized trial in Nantes, has proved to be ineffective in severe vascular IUGR.

Citrulline is a natural aminoacid precursor to arginine and in contrast to L-arginine escapes uptake in the liver and appears directly in the peripheral blood converted by the kidney in arginine, released into the systemic circulation, Citrulline may therefore be more effective in the treatment of pre-eclampsia.

This prospective, randomized, comparative and double-blinded study aims to prolong pregnancy for patients with pre-eclampsia before 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years old
* pregnant woman
* singleton pregnancy
* woman with pre-eclampsia (<36 weeks) without indication of forthcoming extraction
* subjects affiliated with an appropriate social security system
* subjects out of context of guardianship
* written signed informed consent form

Exclusion Criteria:

* age < 18 years old
* isolated hypertension or isolated proteinuria
* severe pre-eclampsia with indication of forthcoming extraction in emergency
* term pregnancy >= 36 Weeks when diagnosis is done
* multiple pregnancy
* lactose intolerance
* context of guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
number of days between the therapeutic initiation and childbirth | childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Nobert Winer, Dr, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - CHU de Nantes, Nantes
  - Hôpital Cochin (Maternité Port-Royal), Paris

REFERENCES:
- [Derived] Winer N, Misbert E, Masson D, Girault A, Alexandre-Gouabau MC, Ducarme G, Dochez V, Thubert T, Boivin M, Ferchaud-Roucher V, Pere M, Darmaun D. Oral citrulline supplementation in pregnancies with preeclampsia: a multicenter, randomized, double-blind clinical trial. Am J Clin Nutr. 2025 Feb;121(2):488-496. doi: 10.1016/j.ajcnut.2024.12.001. Epub 2024 Dec 9. PMID 39638148